CLINICAL TRIAL: NCT07243184
Title: A Prospective, Multicenter Clinical Trial Evaluating the Feasibility and Safety of Polymer Artificial Heart Valve for the Treatment of Mitral Valve Diseases
Brief Title: The Feasibility Study of Polymer Artificial Heart Valve for the Treatment the Mitral Valve Disease.
Acronym: HeartEpoch
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai HeartEpoch Medical Technology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Jiangang Wang, Director of valve and AF surgical center, Beijing Anzhen Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE2025SVMZG01
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Mital Valve Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polymer Artificial Heart Valve (Experimental): Device: Polymer Artificial Heart Valve Mitral valve replacement
  Interventions: Device: mitral valve replacement

INTERVENTIONS:
Device: mitral valve replacement — device: polymer artificial heart valve mitral valve replacement

SUMMARY:
The study aims to evaluate the feasibility and safety of polymer artificial heart valve designed and developed by Shanghai HeartEpoch Medical technology Co. Ltd. for the treatment of the mitral valve diseases.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 60 years old;
2. severe aortic regurgitation or severe aortic stenosis confirmed by ECHO;
3. surgical mitral valve replacement;

Exclusion Criteria:

1. LVEF < 50%;
2. History of cardiac surgery or history of cardiac intervention( within 1 year), Concurrent cardiac surgery(excluding tricuspid valve repair surgery or atrial fibrillation ablation) or cardiac interventional procedures;
3. STS ≥8；
4. intracardiac mass, thrombus or neoplasm confirmed by echo;
5. Coronary artery disease that requires revascularization；
6. A pacemaker need to be implanted;
7. Severe macrovascular lesions require surgical treatment;
8. Patients with active bleeding, bleeding tendencies or those who are unable to receive anticoagulant therapy；
9. There was evidence of acute myocardial infarction within 1 month before the surgery (Q-wave MI or non-Q-wave MI, CK-MB ≥ twice the normal level and/or elevated troponin)；
10. here was a history of cerebrovascular events (CVA) within 1 month before the surgery, including ischemic and hemorrhagic strokes, but excluding transient ischemic attacks (TIA);
11. Confirmed or suspected diagnosis of infective endocarditis or other active infections;
12. There are diseases that significantly affect the evaluation of treatment, such as patients with neurological disorders that affect cognitive abilities, and patients with malignant tumors and an expected lifespan of no more than one year；
13. Other situations in which patients are not suitable to participate in this trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
The composite incidence rate of all-cause mortality and reoperation | 3 months

SECONDARY OUTCOMES:
Implantation success rate | after the operation
The improvement of 6 minutes walk testing(6MWT) from baseline | 3months, 6months
Performance evaluation of implanted valves | 1 day after operation, 7 days after operation, 1 months after operation, 3 months after operation.
The improvement of NYHA from basement | 7 days after operation, 30 days after operation, 3 months after operation